CLINICAL TRIAL: NCT03550339
Title: Regulation of Energy Balance and Metabolism - Mechanisms Behind and Beyond Obesity and Weight Loss
Acronym: BALANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: VTT Technical Research Centre of Finland (Other); Kuopio University Hospital (Other); Alfido Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 327/2016
Record Dates: First submitted 2016-12-19; First posted 2018-06-08 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Obesity; Appetitive Behavior
Keywords: obesity; appetite; food reward; hormonal responses; psychophysiological responses; implicit measures; explicit measures
MeSH Terms: conditions — Obesity; Appetitive Behavior | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SURG (Active Comparator): subjects attending bariatric surgery
  Interventions: Procedure: SURG
- DIET (Active Comparator): subjects attending dietary weight loss program
  Interventions: Behavioral: DIET
- HAES (Active Comparator): subjects attending Health At Every Size weight management program
  Interventions: Behavioral: HAES

INTERVENTIONS:
Procedure: SURG — bariatric surgery according to Finnish Current Care Guidelines for Obesity in adults
  Arms: SURG
Behavioral: DIET — dietary weight loss program according to Finnish Current Care Guidelines for Obesity in adults
  Arms: DIET
Behavioral: HAES — treatment is based on the previously published procedure (e.g. Bacon et al. 2002) and Health At Every Size trademark, consisting of body acceptance, eating behaviour, physical activity, nutrition, and social support
  Arms: HAES

SUMMARY:
The study aims to investigate homeostatic and hedonic mechanisms regulating appetite, energy balance and metabolism in obesity and the effects of three distinct obesity treatments on these regulatory mechanisms.

DETAILED DESCRIPTION:
Obesity is widely acknowledged health problem affecting millions of people globally. Enormous efforts have been made to solve the problem, but long-term results of the conventional weight loss and/or weight management strategies have been poor indicating still inadequate understanding of the problem. Surgical, rather than weight-centred lifestyle interventions, have proved to be the most effective tool available to treat obesity within individuals suitable for obesity surgery. Current surgical interventions are, however, suitable only for a small subset of obese individuals. In general, there is a need for development of new approaches and therapies that are safer and more individualized to each patient in the struggle against obesity and related disorders. To achieve these goals, research must focus to investigate and understand the complex homeostatic and hedonic regulation of eating behavior and energy balance in different physiological and pathological conditions.

This study aims to investigate homeostatic and hedonic mechanisms regulating energy balance and metabolism in obesity and the effects of three distinct obesity treatments on these regulatory mechanisms. The regulatory mechanisms are investigated at the level of metabolism, autonomic and central nervous systems as well as subjective, both implicit and explicit, experiences.

A total of 90 obese female volunteers (18-65 years, body mass index > 35 kg/m2), of which 30 females waiting for bariatric surgery (SURG), 30 females attending a dietary treatment program for obesity (DIET) and 30 females attending Health at Every Size (HAES) program, will participate in the study. The obesity treatment for SURG and DIET groups follows the principles of the Current Care Guidelines for Obesity (adults) and the treatment for the HAES group applies the strategies of the non-diet wellness-based HAES program. The treatment programs of the DIET and HAES groups include 8-10 weekly group sessions organized by authorised nutritionist.

The study includes also two four-hour visits at the research laboratory of the Institute of Public Health and Clinical Nutrition, University of Eastern Finland, the first visit organized before the participants attend any of the obesity treatments and the second visit 12 months later. During the laboratory visits psychophysiological signals (EEG, ANS, facial EMG and eye tracking) are monitored and blood samples taken throughout the experimental period. Participants will also perform two computer-based test sessions, the first one at baseline and the second before a snack meal. Two meals (breakfast and snack meal) are offered to the participants during the experiment in order to study the regulatory mechanisms of interest both at the homeostatic and hedonic states.

ELIGIBILITY:
Inclusion Criteria:

* body mass index >34 kg/m2
* native finnish speaker
* right-handed

Exclusion Criteria:

* pregnancy or breast feeding
* severe visual impairments, severe scalp skin lesions or intracranial bleeding during previous six months
* severe neurological, psychiatric or cardiovascular disease
* type 1 or 2 diabetes mellitus
* use of weight loss medications or other treatments known to affect weight
* heavy alcohol use
* any other condition (medical or other) the principal investigator considers as an obstacle to participation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Implicit associations | Change from baseline D-score at 1 year
  D-score of Implicit Association Test
Explicit ratings | Change from baseline visual analogue scale at 1 year
  Ratings on visual analogue scales for wanting and liking of presented foods

SECONDARY OUTCOMES:
Event-related potentials | Change from baseline event-related potentials at 1 year
  Event-related potentials measured by EEG
Glucose | Change from baseline glucose at 1 year
  Plasma glucose, fasting, postprandial
Insulin | Change from baseline insulin at 1 year
  plasma insulin, fasting, postprandial
Ghrelin | Change from baseline ghrelin at 1 year
  plasma ghrelin, fasting, postprandial
Leptin | Change from baseline leptin at 1 year
  serum leptin, fasting
Peptide YY | Change from baseline PYY at 1 year
  plasma peptide YY, fasting, postprandial
Endocannabinoids | Change from baseline endocannabinoids at 1 year
  plasma endocannabinoids, fasting, postprandial
Weight | Change from baseline weight at 1 year
  body weight, fasting
Eating behaviour | Change from baseline eating behaviour at 1 year
  self-reported questionnaires
Psychosocial characteristics | Change from baseline psychosocial characteristics at 1 year
  self-reported questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Leila J Karhunen, PhD, Principal Investigator — University of Eastern Finland

IPD SHARING:
Plan to Share IPD: No